CLINICAL TRIAL: NCT01113086
Title: Selective Modulation of Cognitive, Affective, and Motor Function by Transcranial Direct Current Stimulation as Co-adjuvant Therapy in Parkinson's Disease.
Brief Title: Use of Noninvasive Brain Stimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2009-P-001806
Record Dates: First submitted 2010-04-20; First posted 2010-04-29 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; Transcranial direct current stimulation; Motor function; Cognitive function; Affective function
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Left active anodal DLPFC (Experimental): We will place the anodal electrode on the left dorsolateral prefrontal cortex. Stimulation will be given at 2 mA for a total of 20 mins for 10 consecutive sessions (Monday through Friday).
  Interventions: Device: Transcranial direct current stimulation
- Right active anodal DLPFC (Experimental): We will place the anodal electrode on the right dorsolateral prefrontal cortex. Stimulation will be given at 2 mA for a total of 20 mins for 10 consecutive sessions (Monday through Friday).
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Placebo Comparator): Sham tDCS: For sham-controlled tDCS subjects, the same montage will be used; however current will be applied for only 30 seconds.
  Interventions: Device: Transcranial direct current stimulation
- Open-Label Arm (Other): In addition to this study we will have an open label arm in which subjects who received sham stimulation through the course of the study will have the opportunity to receive active stimulation free of charge. The same parameters and identical procedures as is done in the original study will be used. Data will be collected as an open label, which will therefore provide additional information. Data obtained from this open label portion of the study will be kept separate.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Subjects will receive a total of 10 stimulation sessions on consecutive days, Monday- Friday for a total of two weeks. During each session, 2 mA of tDCS will be applied for 20 minutes over the left or right DLPFC (active or sham).
  Other Names: tDCS, direct current stimulation

SUMMARY:
The purpose of this research is to determine whether repetitive sessions of transcranial direct current stimulation (tDCS) to the prefrontal cortex can enhance the cognitive, affective and motor functioning of those with Parkinson's Disease.

In this study we will compare active tDCS with sham tDCS. Each subject will receive two consecutive weeks of stimulation (Monday through Friday). A battery of neuropsychological and affective tests will be administered throughout the duration of the study.

DETAILED DESCRIPTION:
Note that this study is a two-center study (the other center is Beth Israel Deaconess Medical Center - PI - Alvaro Pascual-Leone)

* Further study details are provided by Spaulding Rehabilitation Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "probable" PD, defined by the presence of at least 2 out of 3 cardinal motor features of PD (resting tremor, rigidity, and bradykinesia, plus a sustained and significant response to dopaminergic treatment);
* Age 40 or over;
* Taking stable medications for at least 30 days

Exclusion Criteria:

* Features suggestive of other causes of parkinsonism/ parkinson-plus syndromes;
* History of deep brain stimulation or ablation surgery, mass brain lesions;
* History of schizophrenia, schizoaffective disorder, other psychosis, bipolar illness, alcohol/drug abuse within the past year;
* Need for rapid clinical response due to conditions such as initiation, psychosis, or suicidality;
* Contraindications to tDCS*

  * metal in the head
  * implanted brain medical devices
* Unstable medical conditions (eg. uncontrolled diabetes, uncompensated cardiac issues heart failure, pulmonary issues, or chronic obstructive pulmonary disease)
* Pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement in general motor functioning in patients with Parkinson's. | after treatment (10 days) and at follow up (1 and 2 months after final stimulation)
  Measured by various indexes, including Unified Parkinson's Disease Rating Scale (UPDRS), Simple Reaction Time, 4-Choice Reaction Time, Purdue Pegboard Test, Finger tapping, walking time, buttoning up and supination-pronation.

SECONDARY OUTCOMES:
Evidence of improvement in cognitive functioning in the areas of: executive function, reasoning, visuospatial ability, and working memory for patients with Parkinson's. | after treatment (10 days) and at follow up (1 and 2 months after final stimulation)
  Will be measured by The Stroop Test, Hooper Visual Organization Test, Digit Span Test, Trail Making Test B.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Spaulding Rehabilitation Hospital; Ross Zafonte, DO, Study Chair — Spaulding Rehabilitation Hospital
Locations (2):
- United States (2):
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Berenson Allen Center for Noninvasive Brain Stimulation, Boston, Massachusetts